CLINICAL TRIAL: NCT00780832
Title: Comparison of Caffeine Reduction and Anticholinergic Medications for Treatment of Overactive Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient elligible patients available in a reasonable time frame.
Sponsor: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB #4121
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2013-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; dietary caffeine; anticholinergic medication; lifestyle modification; incontinence; urinary frequency
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Caffeine reduction through diet and beverage counselling
  Interventions: Behavioral: Dietary Caffeine reduction
- 2 (Active Comparator): Anticholinergic medication
  Interventions: Drug: Anticholinergic medication

INTERVENTIONS:
Behavioral: Dietary Caffeine reduction — Participants are counseled about reduction of dietary caffeine, given written information and a bladder control log.
  Other Names: Lifestyle modification
  Arms: 1
Drug: Anticholinergic medication — Detrol LA 4mg. orally, once daily for 30 days
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effects of caffeine reduction/elimination on urinary symptoms in women with overactive bladders and compare this therapeutic approach to anticholinergic therapy. We hope to show a reduction in symptoms with caffeine reduction and determine how effective caffeine reduction is compared to medication. If caffeine reduction is shown to be beneficial, women may be encouraged to use this strategy before resorting to medications.

DETAILED DESCRIPTION:
Urinary symptoms such as frequency, urgency, nocturia, and incontinence occur in many women. Overactive bladder (OAB) accounts for forty to seventy percent of urinary incontinence. These symptoms can be mildly annoying to life altering. Many women wear pads or adult diapers daily and avoid social situations for fear of embarrassment. It is felt that up to sixteen percent of the adult population may suffer from these symptoms and many of these women seek medical help.

Currently, the standard of care for OAB includes some combination of lifestyle modification counseling, bladder retraining, or anticholinergic medications. It is anticipated that stimulants such as caffeine irritate the bladder and exacerbate OAB symptoms. There have been a few studies looking at the effect of caffeine but interventions have varied, and the results have been mixed.

Perhaps the most common treatment for significant OAB symptoms is the prescription of anticholinergic medications. We know that these are efficacious in many women but they can be expensive and have significant side effects4. In fact, many women discontinue their anticholinergics due to dry mouth, dry eyes, gastrointestinal, and genitourinary effects.

To date there have been no studies comparing caffeine reduction to anticholinergic medications.

Research Questions

1. Does caffeine reduction decrease OAB symptoms?
2. Does the amount of caffeine consumed relate to symptom severity?
3. If symptoms do improve with caffeine reduction, are women compliant with this treatment?
4. How does caffeine reduction compare to anticholinergic medication in treating OAB?

Study Goal:Compare caffeine reduction to anticholinergic medication as a treatment for overactive bladder.

Study Design:Randomized prospective study. Eligible participants will be randomized to either the anticholinergic arm or the caffeine reduction arm.

ELIGIBILITY:
Inclusion Criteria:

1. Women with OAB symptoms including urgency, frequency (voids ≥8/day), and urge incontinence
2. Women who consume > one cup (250ml) caffeinated beverage per day
3. Women who score $ 6 on the QUID Questionnaire for urgency symptoms

Exclusion Criteria:

1. Women currently receiving treatment for OAB symptoms
2. Women with narrow angle Glaucoma
3. Women taking anticholinergics or loop diuretics
4. Women with an untreated urinary tract infection. After resolution of the UTI, and if all other eligibility criteria are met, the woman can be a candidate for inclusion in the study.
5. Women with a diagnosis of painful bladder syndrome or other abnormal urinary tract lesions
6. Women scoring >4 on the QUID Questionnaire for stress symptoms
7. Women with de novo symptoms following surgery
8. Women with major pelvic prolapse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in Bladder Function Questionnaire score | 30 days

SECONDARY OUTCOMES:
Does the amount of caffeine consumed relate to symptom severity? | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Farrell, MD, FRCSC, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada